CLINICAL TRIAL: NCT02113605
Title: Exposure-Based CBT for Children With Functional Gastrointestinal Disorders - Development of a Protocol
Brief Title: Cognitive Behavior Therapy (CBT) for Children With Functional Gastrointestinal Disorders
Acronym: CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ola Olen, MD, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FGID Child Pilot-0
Record Dates: First submitted 2014-04-01; First posted 2014-04-14 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Functional Gastrointestinal Disorders (FGID); FGID According to the Rome III Criteria; Irritable Bowel Syndrome (IBS); Functional Abdominal Pain; Functional Dyspepsia
Keywords: Functional gastrointestinal disorders; FGID; Recurrent abdominal pain; Abdominal pain; pain-predominant functional gastrointestinal disorders; Pediatric pain
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome; Abdominal Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive behavior therapy (Experimental): All included children are treated with a face-to-face exposure-based cognitive behaviour therapy for 10 weeks. There will be no comparison arm.
  Interventions: Other: Cognitive behavior therapy

INTERVENTIONS:
Other: Cognitive behavior therapy — Exposure-based cognitive behavior therapy in a 10 week face-to-face treatment

SUMMARY:
The purpose of the trial is to develop a treatment protocol to be used in trials studying internet-delivered CBT for children with functional gastrointestinal disorders (FGID). The study size is not based on power calculations but the estimated sample necessary to develop a treatment protocol. This study will include 20-30 children with FGID and their parents who will be treated individually (face-to-face). The treatment consists of 10 weekly sessions of exposure-based CBT. The study uses a pre- post-design with no control group.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8-12 years
* A diagnosis of a functional gastrointestinal disorder by a treating physician

Exclusion Criteria:

* Concurrent serious medical condition or gastrointestinal symptoms likely caused by an organic disorder.
* Psychiatric disorder more urgent to treat than the abdominal pain.
* On-going psychological treatment.
* Absence from school more than 40 %.
* Ongoing maltreatment, violence or severe parental psychiatric illness.
* Pronounced language or learning difficulties that hinder the child to benefit from the treatment.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in Faces Pain Rating Scale (FACES) from baseline to 10 weeks | Baseline and 10 weeks
Change in Faces Pain Rating Scale (FACES) from baseline to 8 months. | Baseline and 8 months.

SECONDARY OUTCOMES:
Change in Gastrointestinal Symptom Rating Scale (GSRS-IBS) from baseline to 10 weeks. | Baseline and 10 weeks.
Change in Children´s Somatization Inventory (CSI 24) from baseline to 10 weeks | Baseline and 10 weeks.
Change in Gastrointestinal Symptom Scale (PedsQL Gastro) from baseline to 10 weeks | Baseline and 10 weeks.
Change in Functional Disability Index (FDI) from baseline to 10 weeks. | Baseline and 10 weeks.
Change in Pain Reactivity Scale from baseline to 10 weeks. | Baseline and 10 weeks.
Change in IBS-behavioral responses questionnaires (IBS-BRQ) from baseline to 10 weeks. | Baseline and 10 weeks.
Change in Spence Children Anxiety Scale (SCAS) from baseline to 10 weeks. | Baseline and 10 weeks.
Change in Child Depression Inventory (CDI) from baseline to 10 weeks. | Baseline and 10 weeks.
Change in Pain Interference Index (PII) from baseline to 10 weeks. | Baseline and 10 weeks.
Change in Pediatric Quality of Life Inventory (Peds QL) from baseline to 10 weeks. | Baseline and 10 weeks.
Change in Gastrointestinal Symptom Rating Scale (GSRS-IBS) from baseline to 8 months. | Baseline and 8 months
Change in Children´s Somatization Inventory (CSI 24) from baseline to 8 months | Baseline and 8 months.
Change in Gastrointestinal Symptom Scale (PedsQL Gastro) from baseline to 8 months. | Baseline and 8 months.
Change in Functional Disability Index (FDI) from baseline to 8 months. | Baseline and 8 months.
Change in IBS-behavioral responses questionnaires (IBS-BRQ) from baseline to 8 months. | Baseline and 8 months.
Change in Spence Children Anxiety Scale (SCAS) from baseline to 8 months. | Baseline and 8 months.
Change in Child Depression Inventory (CDI) from baseline to 8 months. | Baseline and 8 months.
Change in Pain Interference Index (PII) from baseline to 8 months. | Baseline and 8 months.
Change in Pediatric Quality of Life Inventory (Peds QL) from baseline to 8 months. | Baseline and 8 months.
Change in Pain Reactivity Scale from baseline to 8 months. | Baseline and 8 months.

OTHER OUTCOMES:
Change in Parental Behavior FGID (PB-FGID) from baseline to 10 weeks. | Baseline and 10 weeks.
Change in Parental Behavior FGID (PB-FGID) from baseline to 8 months. | Baseline and 8 months.
Change in Adult responses to children´s symptoms (ARCS) from baseline to 10 weeks. | Baseline and 10 weeks.
Change in Adult responses to children´s symptoms (ARCS) from baseline to 8 months. | Baseline and 8 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ola Olén, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Child and Adolescent Psychiatry in Stockholm, Stockholm, Sweden